CLINICAL TRIAL: NCT00245778
Title: fMRI Study of Grasping in Autistic Patients
Status: Terminated | Type: Observational
Why Stopped: All the patients were included
Sponsor: University Hospital, Tours (Other)
Other Study IDs: PHRC-R-2003-INCA
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The aim of the study is to localise brain regions involved in objects recognition, in planification and adjustment of grasping, in prehension with and without eye control. The study is conducted in normal and autistic adults. We hypothesize different activations in these two populations.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of autistic disorder, right-handed, DQ>50

Exclusion Criteria:

* epilepsia, psychotropic drugs

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Barthelemy, MD, PhD, Principal Investigator — University hospital of Tours
Locations (1):
- University hospital of Tours, Tours, France